CLINICAL TRIAL: NCT04634773
Title: Unravelling the Etiology of Shoulder Osteoarthritis
Acronym: UESOA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: University of Ottawa (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 20200766-01H
Record Dates: First submitted 2020-11-12; First posted 2020-11-18 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Osteoarthritis of the Shoulder
Keywords: T1Rho MRI; qCT; Motion Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Early Degeneration ('Disease') (Experimental): Those who have posterior subluxation of the humeral head and show early signs of degeneration in their shoulder.
  Interventions: Radiation: Low-dose CT; Other: T1Rho MRI; Other: Motion Analysis
- Group 2: No Degeneration ('Healthy') (Active Comparator): Those who have posterior subluxation of the humeral head and show no signs of degeneration.
  Interventions: Radiation: Low-dose CT; Other: T1Rho MRI; Other: Motion Analysis

INTERVENTIONS:
Radiation: Low-dose CT — A low-dose, or quantitative (q) CT scan will be performed on the shoulder. This CT scan will be done to assess the bony structure of the shoulder, as well as bone strength, which can influence the health of the cartilage.
  Group 1 participants will complete this scan at baseline, 2-years and 4-years in the affected shoulder, and at baseline and 4-years in the opposite, unaffected shoulder.
  Group 2 participants will complete this scan at baseline, 2-years and 4-years.
Other: T1Rho MRI — A T1Rho MRI will be performed on the shoulder. This imaging technique uses a special sequence and will be used to assess the muscles and tendons around the shoulder.
  Group 1 participants will complete this scan at baseline, 2-years and 4-years in the affected shoulder, and at baseline and 4-years in the opposite, unaffected shoulder.
  Group 2 participants will complete this scan at baseline, 2-years and 4-years.
Other: Motion Analysis — Motion analysis is the study of how joints move and which muscles fire during specific movements. In the lab, participants will be asked to perform movements that they might do during a typical day or when exercising.
  Group 1 participants will complete this scan at baseline, 2-years and 4-years in the affected shoulder, and at baseline and 4-years in the opposite, unaffected shoulder.
  Group 2 participants will complete this scan at baseline, 2-years and 4-years.

SUMMARY:
Osteoarthritis (OA) is a progressive disease resulting from the degradation of synovial joint articular cartilage over time.

The hallmark symptom is diffuse aching and progressive pain made worse with activity. Loss of range of motion and compromised function inevitably follow. This degenerative disease can affect the shoulder joint. When symptoms become refractory to conservative treatment such as anti-inflammatory medication, steroid injections, activity modification or physical therapy; surgery (total or reverse shoulder arthroplasty) may be considered.

Idiopathic shoulder OA is typically characterized by posterior subluxation of the humeral head upon the glenoid and posterior bone loss. An imbalance in the application of forces applied to the proximal humerus by the posterior and anterior rotator cuff muscles has been postulated to be the leading cause of idiopathic shoulder OA. However, there is only preliminary evidence to support this theory and the etiology of this pattern of deformity is unknown. The theory the posterior humeral head subluxation is a precursor to OA is only supported by very low-level evidence and no longitudinal studies have been conducted. As a result, the cause and natural history of shoulder OA remains unknown.

Research into this area is urgently needed to generate knowledge that will inform future treatments aimed at modifying and slowing the progression of shoulder OA and to reduce the need for shoulder replacement therapy.

The aim of this project is to develop an understanding of the pathophysiology of shoulder OA.

DETAILED DESCRIPTION:
Purpose: The aim of this project is to develop an understanding of the pathophysiology of shoulder OA. This project will recruit two groups of 30 participants, (60 participants in total) and follow them over a period of 5-years.

Group 1- Participants with posterior subluxation of the humeral head and show early signs of degeneration in their shoulder 'disease group' Group 2- Participants with posterior subluxation of the humeral head and show no signs of degeneration 'control/healthy' group

Hypotheses: The investigators hypothesize that there are several factors that contribute to the development of shoulder OA. Uncovering those pathways will lead to more targeted therapy. (1) The posterior rotator cuff muscles (infraspinatus/teres minor) apply relatively greater force than the anterior (subscapularis) cuff; an imbalance in the force couple occurs and the humeral head translates posteriorly on the glenoid; progressive posterior subluxation of the humeral head occurs and degeneration of the glenoid and humeral head cartilage follow. (2) Posterior subluxation of the humeral head is associated with progressive cartilage proteoglycan loss. (3) Pre-morbid glenoid morphology including increased retroversion is associated with the development of shoulder OA.

Participant Involvement: The following will be completed with participants: T1Rho Magnetic Resonance Imaging (MRI), quantitative Computed Tomography (qCT), functional and motion analysis at baseline, year 2 and year 4 in the 'affected' shoulder in both groups 1 and 2. These tests will also be conducted on the asymptomatic, contralateral shoulder in Group 1 participants at baseline and year 4. The finite element model validation will be performed in years 2 and 3, and participant-specific finite element analysis (which has no active participant involvement) will occur in years 3 to 5. Overall study analysis will occur in year 5. This project will be done in two-parts. The first part will consist of six participants; assuming further funding is obtained, part two of the study will proceed. The second part of the project will be based on successfully obtaining funds to continue the remainder of the study recruitment (54 participants) and testing. As pilot data is urgently needed to secure granting funds to support this overall project, the investigators will commence with recruiting the first 6 participants. Once further funds are secured, the remaining portion (recruitment of 54 participants) of the project will continue.

Objectives: (1) Determine whether patients with posterior humeral head subluxation have an imbalance between the posterior and anterior rotator cuff muscles. Objective 1 will be assessed through T1Rho MRI, and functional testing/motion analysis.

(2) Determine whether patients with static posterior subluxation of the humeral head are at risk of degenerative changes (i.e. proteoglycan loss). Objective 2 will be assessed through T1Rho MRI and qCT scans.

(3) Determine which joint factors are associated with progression of OA. This will be assessed using qCT scans and finite element model analysis.

Clinical Relevance: The cause is shoulder OA is unknown, and the burden and costs associated with this degenerative disease are increasing with our aging population. Research in this area is urgently needed to generate knowledge which will inform future treatments which may modify and slow the progression of shoulder OA, and to reduce the need for shoulder replacement therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adults <60 years of age
* Posterior humeral head subluxation >55% (determined from imaging)

Exclusion Criteria:

* >60 years of age
* History of shoulder instability
* History of shoulder trauma including fracture
* Neurological disorders of the upper limb
* Imaging evidence of humeral head or glenoid bony deformity
* Rotator cuff pathology
* Labral pathology
* Pre-existing joint deformity (OA) cases greater than grade I (as per Samilson and Prieto)

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-06-23 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
T1Rho MRI | 5-Years Post-Allocation
  MRI will be used to measure the muscle-fat ratio, and tendon thickness. Increased fat-infiltration, and tendon thinning indicates a worse outcome.
qCT (Low Dose CT) | 5-Years Post-Allocation
  Used to measure bone loss and density. Increased bone loss, and decreased density indicate a worse outcome.
Motion Analysis | 5-Years Post-Allocation
  A kinematic evaluation of the shoulder while performing functional tasks will help us determine how the rotator cuff muscle imbalance influences the shoulder joint kinematics.
Finite Element Analysis | 5-Years Post-Allocation
  This will be combined with motion analysis results to gain a better understanding of the internal loading within the tissues of the joint that could explain degenerative changes observed by imaging. Increased stresses, and muscle imbalance result in a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Lapner, MD, FRCSC, Principal Investigator — The Ottawa Hospital Research Institute
Locations (2):
- Canada (2):
  - University of Ottawa, Ottawa, Ontario
  - Carleton University, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: No